CLINICAL TRIAL: NCT06699732
Title: Impact of Mindful Self-Compassion Therapy on Self Harm Behaviors, Emotional Regulation and Quality of Life Among Patients With Borderline Personality Disorder: A Randomized Controlled Trial
Brief Title: Impact of Mindful Self-Compassion Therapy on Self Harm Behaviors, Emotional Regulation and Quality of Life Among Patients With Borderline Personality Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fatima Jinnah Women University (Other)
Responsible Party: Principal Investigator, Asma Mansoor, Principal Investigator, Fatima Jinnah Women University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: FJWU/EC/2024/94
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Psychological Distress; Emotional Regulation; Self Harm; Quality of Life (QOL); Borderline Personality Disorder (BPD)
MeSH Terms: conditions — Emotional Regulation; Self-Injurious Behavior; Borderline Personality Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Who receives intervention i.e. Mindful Self Compassion Therapy
  Interventions: Behavioral: Mindful Self Compassion Therapy
- Waitlist Control (Active Comparator): Who would receive intervention after study completion
  Interventions: Behavioral: Mindful Self Compassion Therapy

INTERVENTIONS:
Behavioral: Mindful Self Compassion Therapy — Mindful Self-Compassion (MSC) therapy is an 8-week program blending mindfulness and self-compassion to improve emotional resilience and well-being.
  Week 1: Introduction - Learn the basics of mindfulness, self-compassion, and reframing self-critical thoughts with kindness.
  Week 2: Mindfulness - Practice observing thoughts and emotions without judgment to build self-awareness.
  Week 3: Self-Kindness - Develop skills to treat yourself with warmth and care during difficult times.
  Week 4: Common Humanity - Explore shared human experiences to reduce feelings of isolation.
  Week 5: Working with Challenges - Learn strategies to respond compassionately to emotional pain.
  Week 6: Growing Compassion - Deepen compassion for yourself and others through guided exercises.
  Week 7: Resilience Building - Strengthen coping skills and foster emotional flexibility.
  Week 8: Integration - Consolidate skills to maintain self-compassion in daily life.

SUMMARY:
The primary purpose of the study is to investigate whether Mindful Self-Compassion (MSC) therapy can significantly reduce self-harm behaviors, improve emotional regulation, and enhance the quality of life in individuals diagnosed with Borderline Personality Disorder (BPD). The study aims to contribute to the existing literature by providing robust evidence on the efficacy of MSC therapy for BPD, which could inform clinical practices and improve treatment outcomes

DETAILED DESCRIPTION:
The current quantitative study will be carried out in two phases. A cross-sectional survey will assess quality of life, emotional regulation, psychological distress, self-harm behaviors, social support, and state of mindfulness during the first phase. A randomized controlled trial (RCT) will be done during the second phase where patients with Borderline Personality Disorder who are identified with psychological distress, low level of social support, and quality of life, will be categorized into two groups i.e. waitlist control group and intervention group through the process of randomization. Then Mindful Self Compassion therapy would be applied to participants in the intervention group. The control group is the waitlist control group so initially no intervention will be given to participants in the control group but the intervention will be given to the control group participants once the study is completed. The Mindful Self Compassion therapy would be implemented on participants using individual and in-person modes. The pre-and post-assessment will be done at Times 1 and 2 within and between control and interventional groups. After doing post-assessment the difference between pre and post-assessment will be compared to explore the efficacy of Mindful Self Compassion Therapy in patients with borderline personality.

ELIGIBILITY:
Inclusion Criteria:

* 1. First time diagnosed non-hospitalized patients of Borderline Personality Disorder.

  2. Patients of Borderline Personality Disorder experiencing psychological distress,low level of quality of life, social support, emotional dysregulation would be included.

  3. Borderline Personality Disorder patients with age 18 years and above (both gender) from outpatient department (OPD) 4. Borderline personality patients who would be able to understand Urdu language and can give the informed consent
* Exclusion criteria

The study would have the following exclusion criteria:

1. Hospitalized patients of Borderline Personality
2. Patients with Borderline Personality having other chronic co-morbid diseases such as cancer, cognitive deficits, and other chronic psychological disorders.
3. Patients with Borderline Personality younger than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-21 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
World Health Organization Quality of Life Scale Urdu Version | 3 months
  It has 26 items and four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains quality of life and general health items. The minimum value is 26 and the maximum value is 130. Higher scores on the scale indicate higher quality of life and low scores indicate low quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Asma Mansoor, PhD Scholar, Principal Investigator — Fatima Jinnah Women University, Rawalpindi, Pakistan
Locations (2):
- Pakistan (2):
  - Commandant Afimh, Rawalpindi, Punjab Province
  - Farid Family Hospital, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No
Due to ethical concerns the data will not be shared. All research findings will be published in aggregate form maintaining patient anonymity

REFERENCES:
- See also: Related Info — https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0248409